CLINICAL TRIAL: NCT04582682
Title: Poly-omic Predictors of Symptom Duration and Recovery for Adolescent Concussion
Status: Active, not recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Steven Hicks, Assistant Professor, Pediatrics, Milton S. Hershey Medical Center
Other Study IDs: STUDY00016155
Record Dates: First submitted 2020-09-24; First posted 2020-10-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-02

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify changes in salivary micro ribonucleic acid (miRNA) levels that are predictive of symptom duration and character following mild traumatic brain injury (mTBI) in children.

DETAILED DESCRIPTION:
The objective of this multi-center study is to refine and validate a saliva RNA assessment for adolescent concussion, yielding a non-invasive test that predicts duration and character of symptoms, and helps guide clinical decisions. To accomplish this goal, the study will enroll 750 adolescents with mTBI. Saliva RNA levels and symptoms will be assessed at <48 hours, 7 days, and 30 days post-injury. Aim 1 will assess the ability of saliva RNA dynamics (Δ from <48 hours to day 7) to predict PPCS 30 days after mTBI (defined by persistence of ≥3 symptoms on day 30, compared with pre-injury state on the Post-Concussion Symptom Inventory; PCSI). RNA accuracy will be compared to a validated clinical prediction tool (5p tool). Aim 2 will assess the ability of saliva RNA dynamics (Δ from <48 hours to day 30) to identify recovered participants on day 30. RNA accuracy will be compared to change in composite score on a standardized reaction time test (from <48hrs to day 30). Completion of these aims will yield an objective biologic test that can be used for prognosis at the time of mTBI, and to aid clinical decisions regarding return-to-learn or return-to-play.

ELIGIBILITY:
Inclusion Criteria:

* Presence of mTBI: defined by criteria from the Berlin Consensus Statement and WHO. Assessment for mTBI status be performed by a licensed clinician per the 2018 CDC guidelines.
* Age at enrollment: 13-18 years of age (inclusive).

Exclusion Criteria:

* > 48 hours after initial mTBI
* Glasgow Coma Scale score of 13 or less
* Previous moderate-to-severe TBI requiring overnight hospitalization
* Unresolved symptoms from previous concussion, or any concussion within the last 3 months
* Abbreviated Injury Scale (AIS) score > 3 (to reduce confounding from poly-trauma)
* Psychiatric illness requiring previous hospitalization;
* Neurological condition (e.g. epilepsy, hydrocephalus) or abnormality on neuroimaging (if performed)
* Intellectual disability that prevents ability to provide informed assent
* Pregnancy
* Active substance use/dependence
* Previous neurosurgery
* Non-fluency in English
* Upper respiratory infection
* Periodontal infection
* Injury to the oropharynx
* Previously enrolled in the same study
* Inability to complete follow-up assessments

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children 13-18 years with mild traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of persistent post-concussive symptoms (PPCS) 30 days after injury | 30 days after injury
  PPCS will be defined by persistence of at least 3 symptoms on day 30, compared with pre-injury state, which will be determined from pre-injury symptoms reported at enrollment using the Post-Concussion Symptom Inventory (PCSI). PCSI is a self reported survey that focus on symptoms in the cognitive, emotional, sleep, and physical domains. This form is called the "Sport Concussion Assessment Tool- 5th Edition" and symptoms are scored from 0 to 6 with 0 being no symptom and 6 being severe. A high score is indicative of a subject experiencing the worst they have experienced this symptom.
Presence or absence of concussion recovery 30 days after injury | 30 days after injury
  Defined as a score of 0 (no difference) on item 22 of the Post-Concussion Symptom Inventory (PCSI); "To what degree do you feel 'differently' than before your injury?" This patient-oriented outcome measure relies on the individual's experience of symptoms to define recovery.PCSI is a self reported survey that focus on symptoms in the cognitive, emotional, sleep, and physical domains. This form is called the "Sport Concussion Assessment Tool- 5th Edition" and symptoms are scored from 0 to 6 with 0 being no symptom and 6 being severe.

SECONDARY OUTCOMES:
Concussion symptom burden and severity | Within 48 hours of injury, 7 days post-injury, and 30 days post-injury
  measured as ranked scores by the PCSI at enrollment, PCSI is a self reported survey that focus on symptoms in the cognitive, emotional, sleep, and physical domains. This form is called the "Sport Concussion Assessment Tool- 5th Edition" and symptoms are scored from 0 to 6 with 0 being no symptom and 6 being severe. Symptom burden will be number of symptoms experiencing and severity will be how sever those symptoms are on the 0-6 scale
Orientation, immediate memory, concentration, and delayed recall performance | Within 48 hours of injury
  measured as ranked scores by the Standardized Assessment of Concussion (SAC) at enrollment, this test scores cognition using orientation (ex. what is todays date), immediate memory (repeating a list of 10 words), concentration (repeating a list of 3-6 numbers backwards and the months of the year backwards), and delayed recall (recalling the list of 10 words from earlier). Subject receives points for each correct answer with lower scores meaning the concussion has affect the subject more
Balance performance | Within 48 hours of injury
  measured by the Balance Error Scoring System (BESS) at enrollment, which includes scoring balance on foam and firm surfaces in three different stances for 20 seconds with eyes closed. One point is give per error. An error is credited to the subject when any of the following occur: moving the hands off of the iliac crests, opening the eyes, step stumble or fall, abduction or flexion of the hip beyond 30, lifting the forefoot or heel off of the testing surface, remaining out of the proper testing position for greater than 5 seconds. The maximum total number of errors for any single condition is 10 with 3 conditions (double leg, single leg and tandem stances) each on each foam and firm surfaces the total maximum BESS score is 60 and the lowest score one can achieve is 0. With 0 being the best and 60 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Hicks, MD, PhD, Principal Investigator — Penn State University, College of Medicine
Locations (5):
- United States (5):
  - Boston Children's Hosptial, Boston, Massachusetts
  - Weill Cornell Medicine/ New York Presbyterian Hospital, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania